CLINICAL TRIAL: NCT02727829
Title: The Assessment of Microcirculation in Brachial Plexus Block Using Perfusion Index and Capillary Filling Time
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, humeyra astan, Resident, Tokat Gaziosmanpasa University
Other Study IDs: 15-KAEK-221
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Circulatory; Change

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: pefusion index measurement — perfusion index measurement using massimo radical 7 device

SUMMARY:
The aim of the present study is to assess the effects of brachial plexus block on microcirculation using pefusion index and capillary filling time.

DETAILED DESCRIPTION:
Microcirculation is very crucial to evaluate the organ function those working properly in human body. The aim of the present study is to assess the effects of brachial plexus block on microcirculation using pefusion index and capillary filling time. A total of 50 patients whose planned to underwent surgery are performed brachial plexus block using ultrasound, and pefusion index, heart rate, blood pressure, capillary filling time are measured at 0, 10th and 20th minutes interval and at postoperative 24th hours. All measures will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score of I and III
* ages between 18 and 70
* upper extremity surgery

Exclusion Criteria:

* not to participate in the study
* reject to perform the intervention
* infection in injection cite
* allergy to local anesthetics
* peripherical vasculary diseases
* psychiatric diseases
* coagulation anomalies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * American Society of Anesthesiologists score of I and III
  * ages between 18 and 70
  * upper extremity surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
perfusion index | five times in one year

SECONDARY OUTCOMES:
capillary filing time | five times in one year
heart rate | five times in one year
blood pressure | five times in one year
oxygen saturation | five times in one year

IPD SHARING:
Plan to Share IPD: No